CLINICAL TRIAL: NCT01824706
Title: A Prospective, Multicenter Observational Study Evaluating the Long Term Safety in Terms of Explantation Rate and Number of Infections of the Custom-made Bioceramic Implant CustomBone™
Brief Title: Prospective, Multicenter Observational Study Evaluating the Long Term Safety of the Custombone Implant
Acronym: CUSTOMBONE
Status: Completed | Type: Observational
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: NT-PMK-1201
Record Dates: First submitted 2013-03-25; First posted 2013-04-05 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Surgery
Keywords: cranial prosthesis
MeSH Terms: interventions — Craniotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- craniectomy: craniectomy
  Interventions: Procedure: craniectomy

INTERVENTIONS:
Procedure: craniectomy — craniectomy

SUMMARY:
A Prospective, Multicenter Observational Study Evaluating the Long Term Safety in Terms of Explantation Rate and Number of Infections of the Custom-made Bioceramic Implant CustomBone™

The patients will be included as soon as they are implanted and follow-up for 2 years. It is observational so no specific exam is planned.

The explantation rate will be measured, that is to say the number of patients whose prosthesis will be removed (with or without any relationship with the implant or the procedure).

ELIGIBILITY:
Inclusion Criteria:

* Patient planning to have a cranioplasty and be implanted with the Custombone™ medical device
* Patient who agrees to take part in the study, or agreement of a representative of the patient in case of patient inability, after being informed by the investigator and having received an information letter

Exclusion criteria:

- Patient who does not accept to take part in the study after being informed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patient implanted with the Custombone prosthesis
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2016-05-01 (Actual)

PRIMARY OUTCOMES:
Explantation rate after 2 years of follow-up | 24 months after implantation
  The main objective of the study is to measure the explantation rate after the implantation of a Custombone TM prosthesis. We will measure the number of patients whose prosthesis has an been removed, with or without any relationship with the implant or the procedure

CONTACTS AND LOCATIONS:
Overall Officials: S Froelich, Principal Investigator — Hospital Lariboisiere Paris
Locations (18):
- France (18):
  - CH Amiens, Amiens
  - CHU Angers, Angers
  - CH de la cote basque, Bayonne
  - CHU la cavale blanche, Brest
  - CHU Beaujon, Clichy
  - CHU Henri Mondor, Créteil
  - CHRU Roger Salengro, Lille
  - CHU Lyon, Lyon
  - CHU Hotel Dieu, Nantes
  - CHU Pasteur, Nice
  - CHU Lariboisière, Paris
  - CHU La¨Pitié Salpêtrière, Paris
  - Hopital Maison Blanche, Reims
  - Hôpital Ponchaillou, Rennes
  - CH Saint Etienne, Saint-Etienne
  - CHU Hautepierre, Strasbourg
  - CH Bretonneau, Tours
  - Clinique du Tonkin, Villeurbanne